CLINICAL TRIAL: NCT01445782
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Inhaled Doses of AZD2115 in Healthy Male Subjects
Brief Title: AZD2115 Multiple Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D3060C00002; Eudract number 2011-002402-75
Record Dates: First submitted 2011-09-27; First posted 2011-10-04 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: Safety; tolerability; healthy; inhaled
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): AZD2115
  Interventions: Drug: AZD2115
- 2 (Placebo Comparator): Placebo to AZD2115
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2115 — Multiple dose, oral inhalation (nebuliser solution)
  Arms: 1
Drug: Placebo — Multiple dose, oral inhalation (nebuliser solution)
  Arms: 2

SUMMARY:
This study will investigate the safety and tolerability of AZD2115 following administration of multiple ascending doses.

DETAILED DESCRIPTION:
A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Inhaled Doses of AZD2115 in Healthy Male Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 45 years with suitable veins for cannulation or repeated venepuncture
* Male subjects should be willing to use barrier contraception ie, condoms and spermicide, from the day of first administration of the AZD2115 until 3 months after administration and must not donate sperm for 3 months after follow-up
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg

Exclusion Criteria:

* Abnormal vital signs, after 10 minutes supine rest, defined as any of the following:

  * Systolic BP >140 mmHg
  * Diastolic BP >90 mmHg
  * Heart rate <40 or >85 bpm
* Prolonged QTcF >450 ms or shortened QTcF <340 ms or family history of long QT syndrome
* Serum potassium concentration of < 3.80 mmol/L on admission (Day -1)
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with the same class to AZD2115 or to excipients
* History or presence of gastrointestinal, pulmonary, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Description of the safety profile in terms of adverse events, blood pressure, pulse, temperature, ECG (Electrocardiogram), lung function (Spirometry), physical examination, safety labs | baseline, up to 30 days
  No formal statistical tests will be performed. Abnormalities will be listed without statistical analysis

SECONDARY OUTCOMES:
Description of the pharmacokinetics (PK) of AZD2115 in terms of area under the curve over the time (AUC) and maximum concentration (Cmax) and terminal half-life | day 1
  PK samples collected post-dose at 5mins, 20mins, 40mins, 1hr, 1.5hrs, 2 hrs, 4hrs, 6hrs, 8hrs, 12hrs, 24hrs 36 hrs, 48hrs
Description of pharmacokinetics (PK) of AZD2115 in terms of Cmax, area under the plasma concentration-time curve from zero to the end of the dosing interval (AUC(0-τ)) | day 17
  PK samples collected post-dose at 5mins, 20mins, 40mins, 1hr, 1.5hrs, 2 hrs, 4hrs, 6hrs, 8hrs, 12hrs, 24hrs 36 hrs, 48hrs 72hrs, 96hrs, 120hrs and 168hrs.
Description of achievement of plasma drug concentration steady state | PK samples collected pre-dose on day 1, day 4, day 6, day 10, day 14, day 17
  An exploratory analysis of achievement of steady state will be evaluated graphically.
Description of pharmacodynamics of AZD2115 in terms of FEV1 (forced expiratory volume in the first second), FVC (forced vital capacity), potassium, glucose, systolic and diastolic blood pressure, pulse rate, heart rate, QTcF | day 1, day 17
  QTcF defined as QT interval corrected for heart rate using Fridericia's formula

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, UK, United Kingdom